CLINICAL TRIAL: NCT05593627
Title: Effect of Lithium Carbonate on Postoperative Sleep and Cognitive Function in Patients Undergoing Heart Valve Surgery With Cardiopulmonary Bypass
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wenfei Tan, Professor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20220920-03
Record Dates: First submitted 2022-10-21; First posted 2022-10-25 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Heart Valve Surgery
Keywords: lithium carbonate; polysomnography
MeSH Terms: interventions — Lithium Carbonate; Tablets; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lithium carbonate (Experimental): Patients undergoing heart valve surgery with cardiopulmonary bypass will take 250mg lithium carbonate .
  Interventions: Drug: Lithium Carbonate 250 MG Oral Tablet
- calcium carbonate (Placebo Comparator): Patients undergoing heart valve surgery with cardiopulmonary bypass will take 500mg calcium carbonate.
  Interventions: Drug: Calcium Carbonate 500 MG Oral Tablet

INTERVENTIONS:
Drug: Lithium Carbonate 250 MG Oral Tablet — Patients undergoing heart valve surgery withcardiopulmonary bypass will take 250mg lithium carbonate
  Arms: lithium carbonate
Drug: Calcium Carbonate 500 MG Oral Tablet — Patients undergoing heart valve surgery withcardiopulmonary bypass will take 500mg calcium carbonate
  Arms: calcium carbonate

SUMMARY:
It has been proved that lithium carbonate can prolong slow wave sleep with few or no side-effects. The aim of the present study is to evaluate postoperative sleep quality of patients undergoing heart valve surgery with cardiopulmonary bypass taken 250mg lithium carbonate after surgery.

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled (randomized, parallel group, concealed allocation), double-blinded trial. All patients undergoing heart valve surgery with cardiopulmonary bypass will be randomized 1:1 to the treatment intervention with lithium carbonate 250mg (Baoqing, Hunan, China) or calcium carbonate 500mg (Reneed, Beijing, China) after surgery. The objective of the trial is to evaluate the lithium carbonate 250mg on the postoperative night sleep quality. Duration of sleep was collected with polysomnography on second postoperative night. (from 20:00pm to 06:00. Mini-Mental State Examination (MMSE) score was performed on the seventh postoperative day

ELIGIBILITY:
Inclusion Criteria:

* Ethnic Chinese;
* Age, 18 to 65 years old;
* Patients undergoing heart valve surgery with cardiopulmonary bypass

Exclusion Criteria:

* Preoperative Pittsburgh Sleep Quality Index global scores higher than 6
* Cognitive difficulties
* Partial or complete gastrectomy
* Previous esophageal surgery
* Previous treated by radiotherapy or surgery
* Inability to conform to the study's requirements
* Body mass index exceeding 30 kg/m2
* Deprivation of a right to decide by an administrative or juridical entity
* Ongoing participation or participation in another study <1 month ago
* Recent (< 3 months prior) use of antibiotics, probiotics, prebiotics, symbiotics, hormonal medication, laxatives, proton pump inhibitors, insulin sensitizers or traditional Chinese medicine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
sleep quality | on the second postoperative night from 20:00 to 6:00
  Duration of sleep was collected with polysomnography on second postoperative night. (from 20:00pm to 06:00am)

SECONDARY OUTCOMES:
serum metabolites | from baseline to postoperative 72 hours
  This study will characterize the serum metabolites of patients before and after heart valve surgery

OTHER OUTCOMES:
Cognitive function | on the seventh postoperative day
  Mini-Mental State Examination (MMSE) score was performed

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided